CLINICAL TRIAL: NCT03146260
Title: Predictors for Successful Sperm Reterival by Testicular Sperm Extraxtion(TESE) in Patients With Non Obstructive Azospermia
Brief Title: TESE and Non Obstructive Azoospermia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Abbass, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB000087987
Record Dates: First submitted 2017-05-06; First posted 2017-05-09 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Azoospermia, Nonobstructive
Keywords: TESE; Sperm retreival; Azoospermia; FSH; LH
MeSH Terms: conditions — Azoospermia, Nonobstructive; Azoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional TESE (Experimental): Conventional testicular sperm extraction (TESE) will be done under anesthesia through small vertical incision in the median raphe, skin, dartos and tunica vaginalis is opened to expose tunica albuginea. The tunica albuginea is incised for about 4mm at the upper pole near the head of epididymis.
  Interventions: Procedure: Conventional TESE
- Microdissection TESE (Experimental): Microdissection testicular sperm extraction (TESE)will be carried under anesthesia micro TESE will be through a transverse incision of the testis covering three-quarters of its circumference, according to a line preserving as much as possible the predominantly transversal sub albugineal vessels. The testis will be opened like a book by gently separating the lobular tissue of both sides. Then, the tissue will be examined under the microscope at ×10-24 magnification to search for areas with dilated whitish tubules, from which numerous microretrievals will be performed.
  Interventions: Procedure: Microdissection TESE

INTERVENTIONS:
Procedure: Conventional TESE — usual procedure for sperm extraction
  Other Names: OrdinaryTESE
  Arms: Conventional TESE
Procedure: Microdissection TESE — Procedure of extraction is performed under the operating microscope
  Other Names: Micro TESE
  Arms: Microdissection TESE

SUMMARY:
Azoospermia is complete absence of sperm in the ejaculate. It accounts for 10-15% of male infertility cases. It is classified as obstructive and non-obstructive azoospermia (NOA). NOA constitutes 60% of all cases of azoospermia. Testicular sperm extraction (TESE) for intracytoplas¬mic sperm injection (ICSI) was first introduced for treatment of obstructive azoospermia in 1993. Soon afterwards testicular sperm were retrieved successfully and used in ICSI in cases of NOA. In the NOA cases, TESE combined with ICSI has been proven to be an acceptable line of treatment. Microdissection TESE may have some theoretical benefits over conventional TESE, but uncertainty exists about its superiority. During a conventional TESE procedure, the testis is exposed through a small incision and one or multiple biopsies are taken blindly. Micro TESE was first introduced in 1999. In this technique, the tunica albuginea is widely opened and examination of the testicular tissue is carried out at 20-25× magnification under an operating microscope allowing visualization of whitish, larger and more opaque tubuli. The concept of this technique is that these tubuli are more likely to contain active spermatogenesis. also no secure clinical predictors of (SR) are demonstrated for both procedures.The recovery of spermatozoa is successful in only 50% of cases and therefore the ability to predict those patients with a high probability of achieving a successful sperm retrieval would be of great value in counselling the patient and his partner . There is no single clinical finding or investigation that can accurately predict the outcome of TESE.An unsuccessful sperm recovery has important emotional and financial implications so objective counselling based on predictive factors may offer realistic expectations for both the couple and physician.

DETAILED DESCRIPTION:
In Assiut university

ELIGIBILITY:
Inclusion Criteria:

* All infertile males with non-obstructive azoospermia

Exclusion Criteria:

* Patient with obstructive azoospermia:

  * Normal FSH
  * Dilated seminal vesicle or ejaculatory duct

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 148 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
prediction model for success of sperm retrieval by TESE in non obstructive azospermic patients | within one hour from the start of the procedure .
  Descriptive statistics for the studied sample will be used as needed. Evaluation of the predictors of sperm retrieval success will be done through a binary logistic regression analysis.

SECONDARY OUTCOMES:
Complications | within three months
  Comparison between conventional TESE and micro TESE as regard complications
sperm retreival rate | within procedure by biological search for sperms in retrieved specimens.
  comparison between two procedures as regard retrieval rate.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa E Abd El moneim, MD, Study Chair — Professor of Urology

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cissen M, Meijerink AM, D'Hauwers KW, Meissner A, van der Weide N, Mochtar MH, de Melker AA, Ramos L, Repping S, Braat DD, Fleischer K, van Wely M. Prediction model for obtaining spermatozoa with testicular sperm extraction in men with non-obstructive azoospermia. Hum Reprod. 2016 Sep;31(9):1934-41. doi: 10.1093/humrep/dew147. Epub 2016 Jul 12. PMID 27406950
- [Background] Abdel Raheem A, Garaffa G, Rushwan N, De Luca F, Zacharakis E, Abdel Raheem T, Freeman A, Serhal P, Harper JC, Ralph D. Testicular histopathology as a predictor of a positive sperm retrieval in men with non-obstructive azoospermia. BJU Int. 2013 Mar;111(3):492-9. doi: 10.1111/j.1464-410X.2012.11203.x. Epub 2012 May 15. PMID 22583840